CLINICAL TRIAL: NCT00698373
Title: Evaluation of Thoracic Tumors With 18F-FMT and 8F-FDG PET-CT: A Clinicopathological Study
Brief Title: Evaluation of Thoracic Tumors With 18F-FMT and 18F-FDG PET-CT A Clinicopathological Study
Status: Completed | Type: Observational
Sponsor: Gunma University (Other)
Collaborators: J~pharma (Industry)
Other Study IDs: Molecular FMT imaging
Record Dates: First submitted 2008-06-12; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Fluorine-18-α-methyltyrosine,; Positron emission tomography,; Fluorine-18-fluorodeoxyglucose,; Lung cancer,
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: PET study

SUMMARY:
L-[3-18F]-α-methyltyrosine (18F-FMT) is an amino-acid tracer for positron emission tomography (PET). The aim of this study was to determine whether PET-CT with 18F-FMT provides additional information for the preoperative diagnostic workup as compared with 18F-FDG PET. Tumor uptake of 18F-FMT was compared with several immunohistochemical markers including L-type amino acid transporter 1 (LAT1).

ELIGIBILITY:
Inclusion Criteria:

* Patients with indeterminate pulmonary nodule suspicious of lung cancer

Exclusion Criteria:

* Patients with other malignancies and those who had received cancer treatment within the past 5 years were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indeterminate pulmonary nodule suspicious of lung cancer were eligible for this prospective study.
Sampling Method: Non-Probability Sample